CLINICAL TRIAL: NCT06891690
Title: Use of TDCS Stimulation in Neurological and Gynaecological Conditions
Acronym: tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20/25
Record Dates: First submitted 2025-02-05; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Spinal Cord Diseases; Nerve Root Disorder; Endometriosis; Dyspareunia; Painful Menstruation; Polycystic Ovary
Keywords: tDCS stimulation; quality of life; pain
MeSH Terms: conditions — Stroke; Spinal Cord Diseases; Radiculopathy; Endometriosis; Dyspareunia; Dysmenorrhea; Polycystic Ovary Syndrome; Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tDCS stimulation (Experimental): The study group will have tDCS stimulation.
  Interventions: Other: tDSC stimulation

INTERVENTIONS:
Other: tDSC stimulation — tDCA stimulation not exceeding 2 mA
  Other Names: tDCS stimulation

SUMMARY:
The aim of the study is to test the effect of tDCS stimulation on upper and lower limb function in neurological patients and to reduce pain in gynaecological patients. And the impact of tDCS stimulation on patients' quality of life. Standardised questionnaires will be used for pre- and post-stimulation evaluation.

DETAILED DESCRIPTION:
Neurological patients:

1. Main objective: The aim of the study is to see whether the use of tDCS stimulation incorporated into a rehabilitation programme in post-stroke patients and patients with spinal cord and nerve root dysfunction following neurosurgery and non-surgery will improve upper and lower limb function.
2. Specific aim: To test whether the application of 1, 5 or 10 tDCS stimulations is sufficient to achieve improvements in upper and lower limb function, taking into account the dominant limb.
3. Description of the study group

   The study will include women and men after stroke and spinal cord and nerve root dysfunction admitted for rehabilitation after surgery and not qualified for surgery, as well as healthy subjects. Study participants will be aged between 20-90 years. Post-stroke subjects with spinal cord and nerve root dysfunction will undergo individual rehabilitation using the PNF (Proprioceptive Neuromuscular Facilitation, Polish for proprioceptive neuromuscular facilitation) neurophysiological method performing upper and lower limb patterns. Rehabilitation will last between one and three months. Inclusion criterion: impairments of upper and lower limb function. Exclusion criterion: no written consent to participate in the study. Due to the assessment to be carried out, participants will be divided into groups:
   * women and men after stroke with and without tDCS stimulation 1, 5 or 10 treatments,
   * women and men with spinal cord and nerve root disorders after surgery with and without tDCS stimulation 1, 5 or 10 treatments,
   * women and men with spinal cord and nerve root disorders not qualified for surgery with tDCS stimulation 1.5 or 10 treatments and without,
   * healthy women and men undergoing all procedures including tDCS stimulation 1.5 or 10 without rehabilitation,
   * women and healthy men undergoing all procedures without tDCS stimulation and rehabilitation.
4. Methods used in the research:

For the purpose of the study to be conducted, the subjects will have an assessment of:

* body weight, body height, body composition using the Tanita BC-418 MA device before the start of the study, the subject stands barefoot on the electrodes in the shape of the foot, in his/her hand he/she also grasps the electrodes while being only in underwear and a measurement is taken, body composition indicators like BMI (Body Mass Index), muscle mass, fat mass, lean body mass and water content will be assessed, measured before the start of the study
* biomechanical and viscoelastic properties of the skin using the MyotonPRO: during the measurement the subject will be in a standing position, the limbs of the subject will be exposed, the skin of both upper limbs (arm and forearm) and lower limbs (thigh and shank) will be assessed, on the anterior, posterior, lateral and medial sides, measurement before and after the test,
* postural stability using the stabilometric platform Coordination, the subject will stand on the platform barefoot only in underwear, upper limbs placed along the torso, measurement will be done with eyes open and closed for a period of 30 seconds, measurement before and after the test,
* upper limb reaction time using the Witty SEM Microgate, taking into account the dominant and non-dominant upper limb, the test person will stand in front of special sensors (semaphores) which will display letters and numbers in different colours, when ready the test person will have to find the small green letter 'a' 20 times as fast as possible. The total time of the test will be counted, the test person will be advised to be in comfortable sportswear (not restricting the movement of the upper limbs), the dominant and non-dominant limbs will be evaluated separately, measuring before and after the test,
* assessment of the squeezing force of the right and left limb (hand dynamometer), test subjects will be asked to grasp the dynamometer and squeeze their hand with maximum force within 5 seconds.
* lower limb reaction time using the Balance Toutor MedTouch platform, the test person will be in comfortable clothing, will be attached by a special harness to the device's extension arm to avoid a possible fall during the test, the test time for one person will last five minutes, the test person will walk on the device's treadmill at a speed of 3 m/s for two minutes, in order to adapt to the walking pace, in front of him/her on a monitor the test subject will see an image of the path in the forest on which he/she is walking in order to divert his/her attention, the device will then elicit a simulated fall reaction in forward, backward and sideways taking into account the test for the dominant and non-dominant lower limb, at the end of the test a record will be obtained for each test subject, recorded by the device in reaction time values, the test will be performed before and after the test,
* tDCS Sooma DUO stimulation, the subject will be subjected to neuromodulation of the motor cortex, the treatment will be carried out in the sitting position, the subject will wear a cap with electrodes attached to the head, the treatment time will be 20-30 minutes, the maximum direct current will be 2 mA, the number of treatments will be 1, 5 or 10 (5 or 10 treatments daily from Monday to Friday) in the afternoon. Before and after the neuromodulation, tests will be carried out for the dominant and non-dominant hand: tapping on a tablet for 30 seconds, reflex flop test on a tablet (there will be glowing points that the subject must touch, the shorter the time to touch all the points, the better the score) and nine-hole peg test. In the course of neurostimulation, after 10 minutes the test person will perform mirror therapy, i.e. The subject will then perform mirror therapy, i.e. movements of the dominant hand controlled in the mirror image (wrist extension - 1 minute and 30 seconds pause, wrist flexion - 1 minute and 30 seconds pause, finger flexion and extension - 1 minute and 30 seconds pause, fist clenching and opening - 1 minute and 30 seconds pause, finger inversion and adduction - 1 minute and 30 seconds pause, middle finger tapping - 1 minute and 30 seconds pause, all fingers tapping - 1 minute).

Completion of questionnaires, the questionnaires used are:

* Roland-Morris disability questionnaire, the questionnaire is completed by the examiner before and after examinations in patients with spinal cord and nerve root disorders,
* Barthel scale, a questionnaire to be filled in by the examiner before and after examinations in stroke patients,
* ASIA scale classification of spinal cord injuries, questionnaire to be filled in by the examiner before and after examinations in patients with spinal cord and nerve root disorders
* Oswestry questionnaire assessment of lumbar spine pain intensity in various activities, questionnaire to be completed by the subject before and after the study,
* Neck Disability Index questionnaire for cervical spine pain before and after the study,
* Sexual Satisfaction Scale for Women (SSS - W - R15), assessment of satisfaction with current sexual life as well as communication with partner and sexual adjustment, questionnaire to be completed by the subject before and after the study,
* male sex life evaluation questionnaire IIEF-5 is filled in by the subject before and after the study,
* Katz scale is filled in by the subject before and after the study,
* Lawton scale is filled in by the subject before and after the study,
* WHOQOL BREF quality of life questionnaire to be completed by the subject before and after the study.

Planned procedures:

1. recruitment of study participants,
2. completion of questionnaires and scales,
3. assessment of weight, height and body composition,
4. ocean biomechanical and viscoelastic properties of the skin using MyotonPRO,
5. assessment of postural stability using the stabilometric platform Coordination,
6. upper limb reaction time using the Witty Sem Macro Gait device taking into account the dominant and non-dominant limb,
7. middle finger tapping test,
8. squeeze strength assessment,
9. lower limb reaction time using the Balance Toutor MedTouch platform,
10. tDCS stimulation.

Gynaecology patients:

1. The aim of the study is to test the effect on pain reduction in women with gynaecological conditions such as endometriosis, painful menstruation, dyspareunia, polycystic ovary syndrome, who have had no treatment other than tDCS stimulation.
2. Specific objective: application of stimulation in quantities; 3 treatments, 5 treatments and 10 treatments.
3. Inclusion criterion: women with selected gynaecological conditions (endometriosis, painful menstruation, dyspareunia, polycystic ovary syndrome) not using any treatment other than tDCS stimulation.

Exclusion criterion: use of treatment other than tDCS stimulation, no written consent to participate in the study.

Patients who do not consent to tDCS stimulation will be placed in the control group.

Gynaecological patients will be asked to complete anonymously standardised questionnaires before and after stimulation, i.e. after 3 or 5 or 10.

Age of female respondents 18-70

For the purpose of the study to be conducted, the subjects will have an assessment of:

body weight, body height, body composition using the Tanita BC-418 MA device before the start of the study, the subject stands barefoot on the electrodes in the shape of the foot, in his/her hand he/she also grasps the electrodes while being only in underwear and a measurement is taken, body composition indicators like BMI (Body Mass Index), muscle mass, fat mass, lean body mass and water content will be assessed, measured before the start of the study biomechanical and viscoelastic properties of the skin using the MyotonPRO: during the measurement the subject will be in a standing position, the limbs of the subject will be exposed, the skin of both upper limbs (arm and forearm) and lower limbs (thigh and shank) will be assessed, on the anterior, posterior, lateral and medial sides, measurement before and after the test,

Standardised questionnaires:

1. quality of life questionnaire WHOQOL-BREF.
2. women's sexual satisfaction scale SSS-W-15 and Female Sexual Function Index
3. Oswestry questionnaire
4. Insomnia Severity Index.

Planned procedures:

1. recruitment of study participants,
2. completion of questionnaires and scales,
3. assessment of weight, height and body composition,
4. assessment of postural stability using the stabilometric platform Coordination,
5. tDCS stimulation. Postural stability using the stabilometric platform Koordynacja, the subject will stand on the platform barefoot in underwear only, upper limbs placed along the torso, measurement will be taken with eyes open and closed for a period of 30 seconds, pre- and post-test measurement, In gynaecological patients of each stimulation is 20 minutes, current intensity to individual patient feeling, not exceeding 2 mA. Stimulation will be performed in a seated position.

Planned use of research results It is planned to present the obtained results in the form of publications in punctuated scientific journals and at Polish and foreign scientific conferences/congresses/symposia. Upon completion of the research experiment, the research participants will receive the results of the research along with their interpretation.

ELIGIBILITY:
Neurological patients

Inclusion Criteria:

* impairment of upper and lower limb function.

Exclusion Criteria:

* no written consent to participate in the study.

Gynaecological patients

Inclusion Criteria:

* women with selected gynaecological conditions (endometriosis, painful menstruation, dyspareunia, polycystic ovary syndrome) with no treatment other than tDCS stimulation.

Exclusion Criteria:

* no written consent to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
body height using Tanita BC-418 MA device | through study completion, an average of 1 year
  height will be measured in centimeters
biomechanical and viscoelastic properties of the skin using MyotonPRO | through study completion, an average of 1 year
  The tissue voltage will be measured in Hertz (Hz)
postural stability using the stabilometric platform Koordynacja | through study completion, an average of 1 year
  the lower the frequency of anterior-posterior and medial-lateral swings, the better the stability
upper limb reaction time using the Witty SEM Microgate device | through study completion, an average of 1 year
  the shorter the time in seconds measured with a stopwatch, the better the result,
assessment of right and left limb compression strength (hand dynamometer) | through study completion, an average of 1 year
  test participants will be asked to grasp the dynamometer and clench their hands at maximum force for 5 seconds, the higher the value measured in kilograms, the greater the hand strength
lower limb reaction time using the Balance Toutor MedTouch platform | through study completion, an average of 1 year
  the shorter the time expressed in seconds, the better the function of the upper limb
tDCS stimulation | through study completion, an average of 1 year
  the subject will be subjected to neuromodulation of the motor cortex, the treatment will be carried out in sitting position, the subject will have a cap on his head with electrodes attached, the treatment time will be 20-30 minutes, the maximum value of direct current will be 2 mA, the number of treatments will be 1, 3, 5 or 10 ( 5 or 10 treatments performed daily from Monday to Friday) in the afternoon
tapping test, reflex Flop test, Nine-Hole-Peg Test | through study completion, an average of 1 year
  before and after the neuromodulation, the shorter the time expressed in seconds, the better the hand performance
questionnaire Rolland-Morris | through study completion, an average of 1 year
  maximum number of points 24, the higher the point value the higher the disability
Barthel scale | through study completion, an average of 1 year
  maximum score 100, the higher the score the more independent the person is
ASIS scale | through study completion, an average of 1 year
  maximum score 5, the higher the score the better the function
Oswestry questionnaire | through study completion, an average of 1 year
  maximum score 50, the higher the score the greater the disability due to lumbosacral pain
Neck Disability Index questionnaire | through study completion, an average of 1 year
  maximum score 50, the higher the score the greater the disability due to cervical pain
Sexual Satisfaction Scale for Women questionnaire | through study completion, an average of 1 year
  Maximum score 55, the lower the score the lower the sexual satisfaction
Female Sexual Function Index questionnaire | through study completion, an average of 1 year
  Maximum score 36, the lower the score the lower the sexual satisfaction
IEF-5 male sex life assessment questionnaire | through study completion, an average of 1 year
  A score of 21 or less may indicate symptoms of penile erectile dysfunction
Katz scale (ADL - Activities of Daily Living) | through study completion, an average of 1 year
  maximum score of 6 indicates preserved activities of daily living, lower scores indicate loss of function
Lawton scale - IADL (basic activities of daily living) | through study completion, an average of 1 year
  The maximum number of points is 27, the lower the score indicates a reduction in everyday functions
WHOQOL-BREF questionnaire | through study completion, an average of 1 year
  130 points (this is the maximum number of points that can be obtained) if it is satisfactory quality of life, 26 points (this is the minimum number of points that can be obtained) if there is no satisfactory quality of life
Insomnia Severity Index | through study completion, an average of 1 year
  maximum score of 28 indicating severity of insomnia symptoms, the lower the score the lower the insomnia symptoms
body weight using Tanita BC-418 MA device | through study completion, an average of 1 year
  body weight will be measured in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- 1Department of Physiotherapy, Poznan University of Physical Education, Faculty of Sport Sciences in Gorzow Wlkp., 61-871 Poznan, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided
When contacted by e-mail, when submitting a publication to a journal, editors often wish to send the raw data.